CLINICAL TRIAL: NCT03117010
Title: A Prospective Cohort for Subjects With Adult Hemophagocytic Lymphohistiocytosis Like Syndrome
Brief Title: Prospective Cohort for Adult Hemophagocytosis
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-08-117
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-11

CONDITIONS: Hemophagocytic Lymphohistiocytoses
Keywords: Hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Steroids; Dexamethasone; Etoposide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 1. Serum sample collection will be done as follows: Baseline, 4 weeks after treatment, Relapse or progression
  2. Germline DNA collection from peripheral blood will be done at the enrollment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophagocytosis: Subjects should fulfill the following criteria
  1. Subjects should have at least one of the following problems
     1. Presence of hemophagocytosis in tissue or bone marrow
     2. Presence of at least 3 conditions among 8 conditions of HLH diagnostic criteria
  2. Age > 18 years
  3. Written informed consents
  Subjects receive steroids and etoposide
  Interventions: Drug: Steroids; Drug: Etoposide

INTERVENTIONS:
Drug: Steroids — High dose dexamethasone 20 mg PO or IV
  Other Names: Dexamethasone
Drug: Etoposide — Etoposide 150mg/BSA

SUMMARY:
This prospective study enrolls subjects who have clinical and laboratory manifestations related with hemophagocytic lymphohistiocytosis. The purpose of the study is to evaluate clinical and biological features of adult hemophagocytic lymphohistiocytosis. The enrolled subjects into this study will be evaluated according to the HLH (hemophagocytic lymphohistiocytosis)criteria and treated with systemic immunosuppressive therapy or chemotherapy. All subjects will be regularly monitored by physicians participating in this study.

DETAILED DESCRIPTION:
Study process is as follows.

1. Informed consent for subjects fulfilling the inclusion criteria.
2. Laboratory evaluation will be done for subjects according to the following diagnostic criteria.

   * Diagnosis will be established if one of either 1 or 2 below is fulfilled

     1. A molecular diagnosis consistent with HLH
     2. Diagnostic criteria for HLH fulfilled (5 out of 8 criteria below)
   * fever ≥ 38.5'C for ≥ 7 days
   * splenomegaly ≥ 3 finger breadth below left subcostal margin
   * cytopenias affecting ≥2 of 3 lineages in peripheral blood (Hemoglobin < 9 g/L, Platelets < 100 × 109/L, Absolute neutrophil count < 1.0 × 109/L)
   * Hypertriglyceridemia and/or hypofibrinogenemia: Fasting triglycerides ≥ 265 mg/dL, fibrinogen ≤ 1.5 g/L
   * Hemophagocytosis in bone marrow or spleen or lymph node
   * Low or absent NK-cell activity (according to local laboratory reference)
   * Ferritin ≥ 500 mcg/L
   * Soluble CD25 (sIL-2 receptor) ≥ 2,400 U/mL

ELIGIBILITY:
Inclusion Criteria:

* Subjects should fulfill the following criteria

  1. Subjects should have at least one of the following problems

     1. Presence of hemophagocytosis in tissue or bone marrow
     2. Presence of at least 3 conditions among 8 conditions of HLH diagnostic criteria
  2. Age > 18 years
  3. Written informed consents

     Exclusion Criteria:
* Subjects cannot satisfy the inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have clinical and laboratory manifestations related with hemophagocytic lymphohistiocytosis.
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Response | 28 days after the 1st treatment
  Response to steroids and etoposide

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Time to date of progression or any kinds of death
Overall survival | 3 years
  Time to date of any kinds of death

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon SE, Eun Y, Huh K, Chung CR, Yoo IY, Cho J, Cho D, Ko YH, Park S, Kim WS, Kim SJ. A comprehensive analysis of adult patients with secondary hemophagocytic lymphohistiocytosis: a prospective cohort study. Ann Hematol. 2020 Sep;99(9):2095-2104. doi: 10.1007/s00277-020-04083-6. Epub 2020 May 21. PMID 32440790